CLINICAL TRIAL: NCT05116969
Title: A Phase 1, Single Dose-Escalation and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous PTX-35 Adminsitration in Healthy Volunteers
Brief Title: A Phase 1 Study of PTX-35 in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew submission to Human Research Ethics Committee as it evaluates the need for healthy volunteer data for development plan.
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: PTX35-101
Record Dates: First submitted 2021-10-20; First posted 2021-11-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Stage 1: PTX-35 Dose Level 1 (Experimental): Dose Level 1: PTX-35 0.1 mg/kg
  Interventions: Drug: PTX-35
- Stage 1: PTX-35 Dose Level 2 (Experimental): Dose Level 2: PTX-35 0.3 mg/kg
  Interventions: Drug: PTX-35
- Stage 1: PTX-35 Dose Level 3 (Experimental): Dose Level 3: PTX-35 1.0 mg/kg
  Interventions: Drug: PTX-35
- Stage 1: PTX-35 Dose Level 4 (Experimental): Dose Level 4: PTX-35 3.0 mg/kg
  Interventions: Drug: PTX-35
- Stage 1: PTX-35 Dose Level 5 (Experimental): Dose Level 5: PTX-35 10.0 mg/kg
  Interventions: Drug: PTX-35
- Stage 2 Multiple Ascending Dose Regimen 6 (Experimental): 4 doses of PTX-35 with each dose separated by 7 days
  Interventions: Drug: PTX-35
- Stage 2 Multiple Ascending Dose Regimen 7 (Experimental): 3 doses of PTX-35 with each dose separated by 14 days
  Interventions: Drug: PTX-35

INTERVENTIONS:
Drug: PTX-35 — PTX-35 is a humanized, affinity matured, IgG2 monoclonal antibody

SUMMARY:
A Phase 1, Single Dose-Escalation and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous PTX-35 Adminsitration in Healthy Volunteers

DETAILED DESCRIPTION:
This is a double blind, placebo controlled, Phase 1 study of PTX-35 administered via IV infusion to healthy male and female participants. This study will be conducted in 2 stages:

* Stage 1 is a single ascending dose (SAD) escalation period in which 5 dose levels of PTX-35 will be evaluated.
* Stage 2 is a multiple dose period in which the highest tolerated dose determined from Stage 1 will be tested in 2 different treatment regimens in 2 cohorts (i.e., 7- and 14- days dosing regimen).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
2. Healthy, male or female volunteers aged 18 to 65 years (inclusive at the time of informed consent).
3. Participants must be in good general health, with no significant medical history, have no clinically significant (CS) abnormalities on physical examination, vital signs, and 12-lead ECG at Screening and/or before administration of the initial dose of study drug.
4. Participants must have a body mass index (BMI) between ≥ 18.00 and ≤ 32.00 kg/m2 at Screening and a total body weight of > 50 kg.
5. Have negative tests for SARS-CoV-2, Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at Screening.
6. Participants must have clinical laboratory values within normal range or abnormal and NCS as specified by the testing laboratory at Screening and admission.
7. Participants must be non-smokers or social smokers who only used nicotine on 5 occasions within 90 days prior to Screening, a negative cotinine test at Screening and Day -1, and ability and willingness to refrain from tobacco products for the duration of the study (from Screening to Follow-up Visit).
8. Participants must have a negative screen for alcohol and DEA Schedule II drugs at Screening and admission.
9. Participants must have no relevant dietary restrictions and be willing to consume standard meals provided.
10. Participants must have good venous access.
11. Females must be not be pregnant and lactating, and must use an acceptable, highly effective double contraception from Screening until study completion, including the Follow-up period unless surgically sterile. Double contraception is defined as a condom AND one other form of the following:

    * Established hormonal contraception (with approved oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones);
    * A vaginal ring or an intrauterine device (IUD);

    Participants that are surgically sterile must have documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner).

    Women not of childbearing potential must be post menopausal for ≥ 12 months. Post menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.

    Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not considered highly effective methods of birth control. Participant complete abstinence for the duration of the study and for 1 month after the last study treatment is acceptable.

    Female participants who are in same-sex relationships are not required to use contraception.

    Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a woman of childbearing potential (WOCBP), the participant and his partner must use an acceptable, highly effective contraceptive method from Screening until study completion, including the Follow-up period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Participants with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.

    WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study.
12. Males must not donate sperm and females must not donate ova for at least 90 days after the last dose of study drug.
13. Participants must have the ability and willingness to attend the necessary visits to the clinical research unit (CRU).

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the Follow-up period.
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant, or presence of respiratory, gastrointestinal, renal, hepatic, hematologic, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
3. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
4. Have a Fridericia's correction factor for QT (QTcF) > 450 ms for male participants and > 470 ms for female participants or history of QT interval prolongation.
5. Have a history of autoimmune disease, hypersensitivity, or cytokine release syndrome (CRS).
6. Have a history of alcoholism or regular alcohol consumption (by self-declaration) at levels which may increase risk of harm from alcohol-related disease or injury; defined as > 10 standard drinks per week (where 1 standard drink = 284 mL of full-strength beer, 30 mL of 40% (alc/vol) spirit, or a 100 mL glass of wine). Participant is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU and for the duration of the study.
7. A history of substance abuse or dependency in the last 12 months, or a history of recreational intravenous drug use over the last 5 years (by self-declaration), or a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, methamphetamines, MDMA, phencyclidine, benzodiazepines, opiates, and cocaine), or alcohol breath test.
8. Have a significant infection or known inflammatory process on Screening or admission.
9. Fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
10. Have acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of Screening or admission.
11. Blood donation or significant blood loss within 60 days prior to the first study drug administration.
12. Plasma donation within 7 days prior to the first study drug administration.
13. History of severe allergic or anaphylactic reactions.
14. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
15. Abnormal ECG findings at Screening that are considered by the Investigator to be CS.
16. History or presence of a condition associated with significant immunosuppression.
17. History of infection that are considered by the Investigator to be life threatening (e.g., meningitis).
18. Infections requiring parenteral antibiotics within the 6 months prior to Screening.
19. Vaccination with a vaccine within the 4 weeks prior to Screening or that is planned within 4 weeks of dosing.
20. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical trial) within the 4 months prior to Screening or 5 half lives, whichever is longer.
21. Alkaline phosphatase (ALP), aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 × upper limit of normal at Screening. Repeat testing at Screening is acceptable for out of range values following approval by the Investigator or delegate.
22. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening.
23. Use of any prescription drugs (other than hormonal contraception; OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD), over the counter (OTC) medication, herbal remedies, supplements or vitamins 2 weeks prior to dosing and during the course of the study without prior approval of the Investigator and MM. Simple analgesia (paracetamol) is permitted (1 therapeutic dose [1 g] per week).
24. Anticipated use of prescription medication or OTC medication during study participation, with the exception of 1 therapeutic dose (1 g) of paracetamol per week and contraceptives.
25. History of surgery or medical intervention, or planned surgery or medical intervention, that could interfere with the objectives of the study or the safety of the volunteer as determined by the Investigator.
26. History of severe allergic reactions (e.g., anaphylaxis) or known sensitivity to any of the constituents of the test product.
27. An employee of the study site or Sponsor who is directly involved in the study, or a family member of such a person.
28. Stage 2 only: Previously participated in Stage 1 of this study.
29. Participant is unwilling to refrain from strenuous exercise (including weight-lifting) from 7 days prior to admission to the CRU until completion of the final Follow-up visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-24 (Estimated); Primary Completion 2022-11-29 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
Primary | Up to 60 days
  To establish the safety number and severity of adverse events of PTX-35 in healthy male and female volunteers